CLINICAL TRIAL: NCT02186704
Title: Sensing Atrial High Rate Episodes With DX System in Implantable Cardioverter Defibrillators Trial
Brief Title: Sensing Atrial High Rate Episodes With Implantable Cardioverter-Defibrillators Trial (The SENSE Trial)
Acronym: SENSE
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1401014661
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Implantable Defibrillators; Implanted Electrodes
MeSH Terms: conditions — Atrial Fibrillation | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ICD with DX system: Implantable cardioverter-defibrillator recipients with DX system
  Interventions: Device: ICD with DX system
- Dual chamber ICD: Dual chamber implantable-cardioverter-defibrillator recipients (retrospective cohort from IMPACT study)
- Single chamber ICD: Single chamber implantable cardioverter-defibrillator recipients (retrospective cohort from Cornell registry)

INTERVENTIONS:
Device: ICD with DX system — Implantable cardioverter defibrillator (ICD) system implantation with single lead with ventricular sensing and pacing and defibrillation combined with dedicated atrial sensing dipole.
  Other Names: Biotronik Ilesto 7 VR-T ICD; Biotronik Lumax Smart S DX ICD lead; Future FDA-approved Biotronik DX-capable ICD and leads
  Groups: ICD with DX system

SUMMARY:
The primary aim of the "Sensing Atrial High Rate Episodes with DX System in Implantable Cardioverter Defibrillators Trial" (SENSE Trial) is to assess the efficacy of a implantable cardioverter-defibrillator (ICD) lead with dedicated atrial sensing dipoles in detecting atrial high rate episodes.

The study hypothesis is that an ICD system with a lead with dedicated atrial sensing dipoles will have a diagnostic yield comparable to that of a standard dual chamber ICD system and superior to that of a standard single chamber ICD system.

DETAILED DESCRIPTION:
The SENSE Trial is designed to study the efficacy of the DX System in detection of atrial high rate episodes (AHREs) in subjects with no prior history of atrial fibrillation. The DX System, or "DX," consists of a Biotronik DX ICD, and the Biotronik Linox Smart S DX lead which is an FDA approved ICD system that incorporates use of an implantable cardioverter-defibrillator (ICD) lead with dedicated atrial sensing dipoles.

The SENSE Trial will be conducted at 8-12 U.S. sites. The lead coordinating site will be at Weill Cornell Medical College. Subjects will be followed for 1 year to assess for the primary endpoints of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills standard indications for ICD implantation
* Subject or legally authorized representative can provide written authorization per institutional requirements
* Subject is intended to be implanted with a complete Biotronik DX system (consisting of a Biotronik Ilesto 7 VR-T DX ICD or any future FDA approved Lumax VR-T DX ICD, and the Biotronik Linox Smart S DX lead), or has been implanted with a complete Biotronik DX system no more than 30 days prior to the date of consent
* Able to comply with Home Monitoring

Exclusion Criteria:

* Subject has prior diagnosis of atrial fibrillation or atrial flutter
* Subject has need for atrial pacing
* Subject unwilling or unable to give informed consent or participate in follow-up
* Subject is unable to comply with Home Monitoring
* Subject is pregnant
* Subject has less than one year estimated life expectancy
* Subject was implanted with a cardiac device capable of detecting AHREs prior to implantation of the Biotronik DX system
* Subject was implanted with Biotronik DX system and had an AHRE detection before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with standard indications for implantable cardioverter-defibrillator implantation and no prior history of atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Atrial High Rate Episode | 1 year
  Atrial high rate episode > 30 seconds in duration

SECONDARY OUTCOMES:
Atrial Sensing (DX System) | 1 year
  P wave amplitudes measured by DX lead system

OTHER OUTCOMES:
Atrial High Rate Episode > 6 Minutes (DX System) | 1 year
  Detection of AHRE > 6 minutes duration by DX lead system

CONTACTS AND LOCATIONS:
Overall Officials: George Thomas, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Massachusetts General Hospital, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - The Ohio State Wexner University Medical Center, Columbus, Ohio
  - Promedica Heart and Vascular Institute, Toledo, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No